CLINICAL TRIAL: NCT00191321
Title: TUHRS Study - Teriparatide Use in Hip Replaced Subjects A Pilot Study on the Use of Teriparatide in Severe Osteoporotic Women With Hip Fracture and Submitted to Hip Replacement
Brief Title: Teriparatide Use in Hip Replaced Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9151; B3D-IT-GHCU
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

INTERVENTIONS:
Drug: Teriparatide

SUMMARY:
A pilot study on the use of Teriparatide in severe osteoporotic women with hip fracture and submitted to hip replacement

The primary objective of this study is to obtain preliminary data, in a pilot group of postmenopausal women with established osteoporosis and a recent hip fracture, who underwent hip replacement 3-6 months before screening phase, about the effect of teriparatide on:

* bone turnover markers: CTx, PINP and BSAP when given at the dose of 20 mcg/day by subcutaneous route for 18 months.

The secondary objectives of the study are as follows:

* Effects of teriparatide on lumbar spine and non-prosthetic femur bone density, as assessed by BMD measurement with dual energy x-ray absorptiometry (DXA)
* Effects of teriparatide on quality of life and back pain during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory postmenopausal women with established osteoporosis, based on the disease diagnostic criteria
2. Presence of more than 1 clinical and/or radiological vertebral fractures OR more than 1 non-vertebral fracture
3. Presence of hip fracture with hip replacement surgical procedure (both uncemented or cemented total hip arthroplastics or endoprosthesis) in the 3-6 months before screening phase
4. Age range 55-85 years
5. Normal or clinically insignificant abnormal laboratory values (as determined by the investigator) including serum calcium, PTH(1 84), and 25 hydroxyvitamin D concentrations, and alkaline phosphatase activity.

Exclusion Criteria:

1. History of diseases which affect bone metabolism, other than primary postmenopausal osteoporosis, such as Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis (included glucocorticoid-induced osteoporosis), hypoparathyroidism, hyperparathyroidism, hyperthyroidism
2. Actual cancer disease or history of malignant neoplasms in the 5 years prior to Visit 2, with the exception of superficial basal cell or squamous cell carcinomas of the skin that have been definitively treated. Subjects with carcinoma in situ of the uterine cervix treated definitively more than 1 year prior to entry into the study may be enrolled.
3. Increased baseline risk of osteosarcoma: Paget's disease of the bone or unexplained elevations of alkaline phosphatase; Prior radiation therapy involving the skeleton
4. Significantly impaired renal function
5. Significantly impaired hepatic function

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Effect of Teriparatide (20 mcg/day for 18 months ) on bone turnover markers: CTx, PINP and BSAP

SECONDARY OUTCOMES:
Effects of teriparatide on lumbar spine and non-prosthetic femur bone density, as assessed by BMD measurement with dual energy x-ray absorptiometry (DXA)
Effects of teriparatide on quality of life and back pain during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- Italy (11):
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alghero
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palermo
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pietra Ligure
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Treviglio
  - For additional information regarding investigative sites for thsi trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine